CLINICAL TRIAL: NCT03334162
Title: Playful Sensorimotor Training to Reduce the Symptoms of Chemotherapy-induced Peripheral Neuropathy in Pediatric Brain Tumor Patients- a Randomized Controlled Trial
Brief Title: Playful Sensorimotor Training in Pediatric Brain Tumor Patients
Acronym: RESET
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: study temporarily paused due to an Amendment request
Sponsor: University of Basel (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dr. Fiona Streckmann, Principal Investigator, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RESET-study
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Cancer; Pediatric Brain Tumor; Chemotherapy-induced Peripheral Neuropathy; Sensorimotor Polyneuropathy
Keywords: Children; Adolescents; Cancer; brain Tumor; exercise; Chemotherapy-induced Peripheral Neuropathy; CIPN; Sensorimotor Training
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This pilot study will follow a prospective, two-armed, randomized controlled design (RCT with follow-up)
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators dealing with the assessments (neurological and sport scientific) and data are blinded, solely the patient as well as the training staff can't be blinded due to the nature of an exercise interventional study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will perform a standardized, age-adjusted, specific playful sensorimotor training (SMT) program twice a week for 12 weeks in addition to usual care.
  Interventions: Behavioral: Sensorimotor training
- Control group (No Intervention): Children in the control group will receive treatment as usual. The control group will be given the opportunity to participate in the intervention after study completion

INTERVENTIONS:
Behavioral: Sensorimotor training — Supervised training sessions will last for about 20 to 30 minutes in total, including a child-specific warm-up and cool-down. The children will be asked to maintain balance in a previously acquired "short-foot-position", knees slightly flexed (30°), without shoes. Training will consist of 5 playful balance exercises, chosen from a standardized pool of exercises according to the child's age, with increasing difficulty (5 degrees of difficulty - e.g. by reducing the base of support, or dual task exercises - per exercise depending on the age group) in order to allow for individual, optimal progression. Each of the 5 exercises will contain of 5 repetitions for 10sec. allowing for a 20sec. rest in between each set and a 1min rest between each exercise in order to avoid neural fatigue. Children will be given a training manual and diary to train at home after the study. Guardians will be instructed in order to be able to assist their children
  Other Names: There are no other intervention names.
  Arms: Intervention group

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a highly prevalent and clinically relevant side-effect of cancer treatment. The severe symptoms such as loss of sensation, numbness, pain, absent reflexes or loss of balance control not only diminish children's quality of life but also affect the medical therapy. To date, there are no effective treatment options to reduce the symptoms of CIPN. Promising results have so far been achieved with specific exercise interventions.

The investigators would therefore like to conduct a prospective, multicenter, two-armed trial (RCT with follow-up). Patients (N=20) will be recruited from the Hospital for Children and Adolescents, Kantonsspital Aarau. Prior to randomization, all primarily eligible patients that have received a platin derivate or vinca-alkaloid, will be screened for symptoms of CIPN. Eligible patients with a neurologically confirmed CIPN will then be randomized either into an intervention group or a control group (CG). Patients in the intervention group will perform a standardized, age-adjusted, specific playful sensorimotor training (SMT) program twice a week for 12 weeks in addition to usual care, while the control group receives treatment as usual. The CG will be given the opportunity to participate in the intervention after study completion. Data change will be assessed at 3 time points: At baseline (T0), after 12 weeks (post intervention testing, T1), and after 12 weeks of follow-up (T2). Primary endpoint is the Ped-mTNS score in order to subjectively as well as objectively assess the severity of CIPN symptoms. It contains a short questionnaire as well as more objective parameters such as light touch sensation, pin sensibility, vibration sensibility, deep tendon reflexes and muscular strength. Additionally, the CIPN symptom pattern will be assessed via nerve conduction studies, CIPN related pain, dorsiflexion and knee extension as well as postural control. Furthermore, investigators will be evaluating patients' level of physical activity, walk to run transition time, lower limb power as well as patients integration in physical education (PE) in school and sport club activities. The investigators hypothesize that patients in the intervention group will be able to reduce relevant symptoms of CIPN, improving related physical functions and enhancing children's social reintegration.

ELIGIBILITY:
Inclusion Criteria:

* patients with a central nervous system (CNS) tumor
* age: ≥ 6 and ≤ 18 years
* neurotoxic chemotherapy treatment is completed 3 months to 2 years ago
* neurotoxic chemotherapy comprised a platinum-derivate or vinca-alkaloid (low grade gliomas: vincristine/carboplatin or vinblastin mono and embryonal tumors as well as ependymomas: cisplatin/ lomustine and vincristine or cyclophosphamide/ carboplatin/ vincristine/ etoposide)

Exclusion Criteria:

* neuropathies of other cause (e.g. diabetes)
* disabilities
* lack of German language that prevent the understanding of the informed consent as well as the instructions for training

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Ped-mTNS score (assesses the change in the severity of CIPN symptoms) | Delta of Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  The Ped-mTNS Score comprises the patient reported outcome, in accordance with pharmaceutical studies to reduce the symptoms of CIPN as well as an objective clinical test battery, resulting in an overall score. The questionnaire contains questions regarding sensory, functional and autonomic symptoms of CIPN and will be used to document and assess the severity of the subjective peripheral neuropathy (PNP) symptoms. The clinical test battery contains light touch sensation, evaluated with Semmes-Weinstein-monofilaments, pin sensibility (MediPin), vibration sensibility assessed with a biothesiometer, deep tendon reflexes of Achilles and patellar tendons and muscular strength examined by a manual muscle test.

SECONDARY OUTCOMES:
short clinical test battery for CIPN | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  The short clinical test battery contains the Achilles- and patella-tendon reflexes assessed with a Taylor reflex hammer, peripheral deep sensitivity assessed with a tuning fork, proprioception with a filament, sense of position by the investigator changing the position of the patients toe and lower leg strength (see knee extension)
Postural control | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  A force plate (Leonardo, Novotec, Pforzheim, Germany) will be used to assess changes in the center of pressure during upright static and dynamic stance. The assessment follows a standardized protocol.
Dorsiflexion function | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  Ankle dorsiflexion strength and active ankle range of motion are measured using a hand-held dynamometer (Alluris, Freiburg, Germany) and a goniometer (Lafayette extendable goniometer), respectively. For measuring ankle dorsiflexion strength, participants are lying in a supine position; legs straight and foot maximal dorsiflexed. The responsible researcher places the dynamometer on the participant's inset of the foot and incrementally increases the force until the patient gives away (break technique). For measuring active ankle range of motion, two measurements are conducted; (1) children are sitting with straight legs (2) children are lying in a supine position with the legs supported by an adequate padding and the knees flexed to minimize potential impact of the flexibility of the gastrocnemius muscle. All dorsiflexion function measurements are carried out bilaterally and repeated two times, recording the best value of each foot as well as a mean value of both feet for analysis.
Knee extension strength | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  In addition to ankle dorsiflexion strength, we will additionally assess knee extension strength to get a better overview of lower leg strength. To measure knee extension strength, a hand-held dynamometer (Alluris, Freiburg, Germany) and the break technique are used, as described in the section "dorsiflexion function". Participants sit upright with a hip and knee angle of 90°.
lower limb power | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  Power and strength of the lower limbs are crucial for any kind of locomotor performance in daily life as well as sports participation. The countermovement jump test is a simple, functional, valid and highly reliable measurement of lower body power that is influenced by sensorimotor training. Following instruction and familiarization trials, children perform 5 consecutive countermovement jumps (CMJ) on a force-plate (Leonardo, Novotec, Pforzheim, Germany). The jumps are performed in an upright position with arms placed akimbo. The applied sampling frequency is 1000 Hz. Jumping height is computed using the flight time method. The best of the five attempts will be analyzed. Between jumps, a break of one minute will be provided.
Walk to run transition time: | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  Fast walking demands a high intramuscular coordination and stability. People with decreased stability and coordination tend to transit from slow walking straight to running as this requires less strength and coordination. The walk-to-run-transition time is the preferred speed at which human change gait from walking to running and is defined as the initial moment where both feet are off the ground at the same time. To assess the participants' preferred walk-to-run-transition time, a treadmill test is performed. After a short familiarization on the treadmill (walking at various speeds), the test protocol provides an age-specific start-speed which is incrementally increased (every 10 seconds by 0,045 m/sec) by the researcher until the participant switches to a run for the first time.
CIPN-related pain | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  In line with pharmaceutical studies to reduce the symptoms of CIPN, we will also measure intensity of CIPN-related pain using a FacesPain scale for children up to 12 years and a visual analogue scale (VAS) for children and adolescents aged 13 or older, both, starting at 0 = no pain, up to 10 = unbearable pain. These measurements have been reviewed and are recommended through the pediatric initiative on methods, measurement, and pain assessment in clinical trials (PedIMMPACT) group.
Participation in PE as well exercise-related leisure activities | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  We would furthermore like to add questions concerning childrens' integration and participation in PE in school as well as in physically demanding leisure activities. For this purpose, children will answer the standardized questionnaire of the KiGGS study (German Health Interviews and Examination Survey for Children and Adolescents) (Bös 2009), offered in two different versions (for kindergartners and for students). Cancer- and treatment-related questions about potential barriers preventing from taking part in sporting activities are added (i.e. anxiety, prohibition by physician or parents or others, lack of time). All questions are answered via interview.
Priority of side-effects | Data will be assessed at 3 time points: At baseline (T0), post assessment after 12 weeks of intervention (T1) and after 12 weeks of follow-up (T2).
  To assess the significance of CIPN, we would like to add a self-developed questionnaire regarding childrens' and parents' prioritization regarding the side-effects of chemotherapy. Therefore, typical CIPN symptoms, further side-effects of chemotherapy as well as their impact on the active lifestyle are described in age-appropriate language; subjective perception and perceived burden can be assessed on a five point-likert scale, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Streckmann, Principal Investigator — University of Basel, Departement of Sport, Exercise and Health
Locations (1):
- Kantonspital Aarau, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No